CLINICAL TRIAL: NCT02708758
Title: Efficacy of Treatment in Women With Gestational Diabetes Mellitus Diagnosed by One Altered Value by the International Association of Diabetes and Pregnancy Study Groups Criteria (IADPSG).
Brief Title: Efficacy of Treatment for Gestational Diabetes Diagnosed by the IADPSG Criteria.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes (Other Government)
Responsible Party: Principal Investigator, ENRIQUE REYES-Munoz MD, Researcher in Medical Sciences, Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONACYT 233634; 212250-3402-10102-02-14 (Registry Identifier: Instituto Nacional de Perinatología, (INPer))
Record Dates: First submitted 2016-02-22; First posted 2016-03-15 (Estimated); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Active Comparator): Medical nutrition therapy plus self monitoring capillary glucose levels and if necessary drug therapy (metformin or insulin) when goals are not met.
  Interventions: Behavioral: Medical Nutrition Therapy
- Routine care group (No Intervention): Prenatal routine care without medical nutrition therapy and without self monitoring capillary glucose levels and drug therapy specific for GDM.

INTERVENTIONS:
Behavioral: Medical Nutrition Therapy — individualized medical nutrition therapy from a qualified nutritionist which took into consideration a woman's pre-pregnancy weight, activity level, dietary intake and weight gain, instructions on how to self- monitoring capillary glucose levels two to four times daily until the levels had been in the recommended range (fasting glucose levels no more than 95 mg/dL and 1 hour postprandial less than 140 mg/dL). Drug therapy will begin with metformin or insulin when capillary glucose levels are not met the recommended levels after at least two weeks of treatment.
  Arms: Treatment group

SUMMARY:
There is a lack of international uniformity in the approach to the screening and diagnosis of gestational diabetes mellitus (GDM). The new diagnostic criteria by the International Association of Diabetes and Pregnancy Study Groups (IADPSG) based on data from the study of Hyperglycemia and Adverse Pregnancy Outcomes (HAPO) have created controversy because of the lack of clinical evidence of treatment benefit for mild GDM and the treatment effects on perinatal outcomes. The purpose of the present study is to know the efficacy of treatment to reduce adverse pregnancy outcomes in Mexican women diagnosed with GDM by IADPSG criteria.

DETAILED DESCRIPTION:
Currently no evidence from randomized clinical trials on the efficacy of treatment of gestational diabetes mellitus (GDM), diagnosed by a single altered value during a 75g oral glucose tolerance test (75g OGTT), proposed by the International Association of Diabetes and Pregnancy Study Groups (IADPSG) to reduce adverse perinatal outcomes (APO). In our institution GDM diagnosis is established with two or more altered values during 75g OGTT, women with one altered value during OGTT are not considered GDM and therefore those women do not receive specific treatment for GDM. We conduct an open randomized clinical trial, two groups, Group 1 (women with treatment for GDM) and group 2 (women with routine care). The diagnosis of GDM will be perform with a single altered value during 75g OGTT: fasting ≥ 92mg / dL, 1-hour ≥ 180 mg / dL and 2-hours ≥ 153 mg / dL. Treatment consist of medical nutritional therapy (MNT), which includes restricted diet 45% carbohydrate, exercise and self-monitoring of glucose, if not reach therapeutic goals metformin and / or insulin will be added.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy between 18-30 week´s gestation
* 75-g oral glucose-tolerance test at 20-30 week´s gestation with only one altered value between: Fasting 92-99 mg/dL

  1. hour 180-211 mg/dL
  2. hour 153-177 mg/dL

     Exclusion Criteria:
* Pregestational diabetes (first diagnosed in pregnancy) defined by altered values during 75-g oral glucose-tolerance test above:

Fasting >126 mg/dL 2 hour >200 mg/dL

-Two or more altered values during oral glucose tolerance test above: Fasting 92 mg/dL

1. hour 180 mg/dL
2. hour 153 mg/dL

   * Multiple pregnancy
   * Active chronic systemic disease as hyperthyroidism, hearth, hepatic or renal disease, immunological disease as lupus and chronic hypertension

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
incidence of large for gestational age | obstetrical resolution (birth)
  Sex specific birth weight for gestational age above the 90th percentile of Mexican fetal growth curves.

SECONDARY OUTCOMES:
incidence of preeclampsia | from 20 weeks of gestation to birth
  incidence of women at fina of gestation that have high blood pressure > 140/90 and proteinuria (more than 300 mg/dl) after 20 weeks of gestation.
incidence of cesarean section | from 26 weeks of gestation to birth
  Extraction of the fetus by means of abdominal hysterotomy.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Reyes-Muñoz, MD, PhD., Principal Investigator — Department of Endocrinology (INPer)
Locations (1):
- Instituto Nacional de Perinatología Isidro Espinosa de los Reyes, Mexico City, Mexico